CLINICAL TRIAL: NCT03979287
Title: Efficacy of a Interferential Current and Therapeutic Exercise Program in Subjects With Chronic Neck Pain
Brief Title: Interferential Current and Therapeutic Exercise Program in Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Alberto Marcos Heredia-Rizo, Assistant Professor, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IFC Therapy and Exercise
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Neck Pain
Keywords: Chronic Neck Pain; Interferential Current Electrotherapy; Therapeutic Exercise; Physical Therapy
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IFC and Therapeutic Exercise Program (Experimental): Patients will receive 10 sessions for two weeks. The duration of each session will be of approximately one hour. Participants will receive treatment with Interferential current therapy plus a program of therapeutic exercise focused on the neck region
  Interventions: Other: Interferential Current and Therapeutic Exercise Program
- Therapeutic Exercise Program (Active Comparator): Patients will receive 10 sessions for two weeks. The duration of each session will be of approximately one hour.This group will only receive the same therapeutic exercise program.
  Interventions: Other: Therapeutic Exercise Program

INTERVENTIONS:
Other: Interferential Current and Therapeutic Exercise Program — The Interferential Current Program will be based on a bipolar application using the Sonopuls 692 device (Enraf Nonius, Rotterdam, The Netherlands). The current parameters will be: a) 4000Hz carrier frequency; and b) 60 Hz AMF with a modulation frequency of 90 Hz. The intensity of the current will be adapted to the sensitivity of each patient.
  The Therapeutic Exercise Program will be applied by a physiotherapist and will consist of:
  1. Ergonomic advices on reducing repetitive movements and/or maintained positions
  2. A protocol of active physiotherapy for neck and shoulder muscles. This protocol will include: active stretching exercises; isometric muscle strengthening exercises; reeducation of the ocular and neck muscles with control retraining exercises
  Arms: IFC and Therapeutic Exercise Program
Other: Therapeutic Exercise Program — The Therapeutic Exercise Program will be applied by a physiotherapist and will consist of:
  1. Ergonomic advices on reducing repetitive movements and/or maintained positions
  2. A protocol of active physiotherapy for neck and shoulder muscles. This protocol will include: active stretching exercises; isometric muscle strengthening exercises; reeducation of the ocular and neck muscles with control retraining exercises
  Arms: Therapeutic Exercise Program

SUMMARY:
Objectives: To analyze the number of sessions needed to achieve a positive impact after combining interferential current therapy and therapeutic exercise, compared with therapeutic exercise alone, on self-reported pain, disability and range of motion in subjects with chronic neck pain.

Design: A randomized, single-blind, controlled trial. Subjects: Patients between 18 and 65 years old, with idiopathic chronic neck pain.

Methods: The experimental group who will perform a combined treatment using Interferential current therapy and therapeutic exercise for two weeks. The control group will receive the same program of therapeutic exercise during the same period of time.

ELIGIBILITY:
Inclusion Criteria:

* Nonspecific mechanical neck pain (chronic neck pain diagnosed by a physician)
* Age between 18 and 65 years old
* Both males and females
* Non apprehension to electrotherapy (determined by the Personal Psychological Apprehension scale- EAPP)
* Self-reported pain higher than 2 in the 11-point Numeric Pain Rating Scale

Exclusion Criteria:

* Metallic implants in the vertebral column
* Apprehension to electrotherapy (a score >45 points in EAPP)
* Cervicogenic headache
* Cervicogenic Dizziness
* Neck pain associated with neurological deficits
* Unexplained fever
* Cervical surgery associated to persistent pain
* Specific diagnostics (cervical myelopathy, cervical stenosis, osteomyopathy)
* Other diagnostics such as visceral pain referred to the neck or non-cervical cause.
* Involvement in litigation
* Manual treatment for the neck-shoulder area in the last month before data collection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-07-13 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Neck pain intensity | From baseline to immediately after treatment
  Participants will rate the intensity of their neck pain at rest on an 11-point numeric pain rating scale, where 0 is no pain and 11 maximum pain. The subjects will be ask to indicate the pain levels that they experienced before treatment and after treatment.
Disability | From baseline to immediately after treatment
  The Neck Disability Index (NDI) will be used in the Spanish version to measure level of disability of the neck area during the daily life activities.
  where under 9 denotes No Disability; from 10 to 29 denotes Slight Disability; from 30 to 49 denotes Moderate Disability; from 50 to 69 denotes Severe Disability and more tan 70 denote Complete Disability.

SECONDARY OUTCOMES:
Range of movement (ROM) | From baseline to immediately after treatment
  The secondary outcome measure will be the active cervical range of motion assessed with the CROM device (Performance Attainment Associates, Lindstrom, MN). The measurements will be made separately for each direction and in a standard sequence: flexion, extension, right lateral flexion, left lateral flexion, right rotation and left rotation. Two measurements will be recorded for each movement and the average of the two measurements will be used in the analysis of results

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Heredia-Rizo, PhD, Study Director — Physiotherapy Department, University of Seville, spain
Locations (1):
- University of Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: No